CLINICAL TRIAL: NCT05051813
Title: The Heidelberg Engineering ANTERION Corneal Epithelium Thickness Precision and Agreement Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2020-1
Record Dates: First submitted 2021-09-08; First posted 2021-09-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Normal Cornea; Corneal Abnormality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal Cornea: 3 repeat measurements on each of the 3 investigational and 3 reference devices
  Interventions: Device: ANTERION
- Corneal Abnormality: 3 repeat measurements on each of the 3 investigational and 3 reference devices
  Interventions: Device: ANTERION

INTERVENTIONS:
Device: ANTERION — 3 repeat measurements on each of the 3 ANTERION devices and 3 reference devices.

SUMMARY:
This is a prospective clinical study that will be conducted at one clinical site located in the United States to assess corneal epithelial thickness parameters with the ANTERION

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 22 years of age
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. With at least one of the following eye status for the corresponding eye population:

   * Normal Cornea
   * Abnormal Cornea: eye with at least one of the following

     a) Keratoconus b) Contact Lens Wearer c) Status Post-Keratorefractive Surgery (at least 30 days between imaging and Keratorefractive Surgery) d) Dry Eye Disease

Exclusion Criteria:

* Exclusion Criteria General

  1. Active infection in either eye
  2. Insufficient corneal reflex, in the study eye
  3. Physical inability to be properly positioned at the study devices or eye exam equipment
* Exclusion Criteria Normal Cornea Group

  4. Abnormal cornea shape or corneal surgery in the study eye

  5. Contact lens wear within 3 months prior to imaging in the study eye

  6. Dry eye disease in the study eye
* Exclusion Criteria Abnormal Cornea Group

  4. For Keratoconus (a):
  * Contact lenses worn within one hour prior to imaging

    5. For Contact Lens Wearer (b):
  * Keratoconus
  * Post-Keratorefractive surgery
  * Contact lenses worn within one hour prior to imaging

    6. For Post-Keratorefractive Surgery (c):
  * Keratoconus
  * Contact lens wear within 3 months prior to imaging in the study eye

    7. For Dry Eye Disease (d):
  * Keratoconus
  * Post-Keratorefractive surgery
  * Contact lens wear within 3 months prior to imaging in the study eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal and Abnormal Cornea populations
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Corneal Epithelial Thickness 0-2mm ring | Through study completion, an average of 1 day
  Reproducibility, repeatability and agreement of Corneal Epithelial Thickness parameters (0-2mm ring) of ANTERION and the reference device
Corneal Epithelial Thickness 2-5mm ring | Through study completion, an average of 1 day
  Reproducibility, repeatability and agreement of Corneal Epithelial Thickness parameters (2-5mm ring) of ANTERION and the reference device
Corneal Epithelial Thickness 5-7mm ring | Through study completion, an average of 1 day
  Reproducibility, repeatability and agreement of Corneal Epithelial Thickness parameters (2-5mm ring) of ANTERION and the reference device
Minimum Thickness from 7mm zone | Through study completion, an average of 1 day
  Reproducibility and repeatability of minimum thickness (7mm zone) of ANTERION and the reference device
Maximum Thickness from 7mm zone | Through study completion, an average of 1 day
  Reproducibility and repeatability of maximum thickness (7mm zone) of ANTERION and the reference device

SECONDARY OUTCOMES:
Adverse Events Rate | Through study completion, an average of 1 day
  Adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischer, MD, Principal Investigator — Fischerr Laser Eye Center, MN, USA
Locations (1):
- Fischer Laser Eye Center, Minneapolis, Minnesota, United States